CLINICAL TRIAL: NCT03402776
Title: Impact of a Fourth Hexavalent Vaccine Dose During Primary Vaccination After Haematopoietic Stem Cell Transplantation
Brief Title: Impact of a Fourth Hexavalent Vaccine After Hematopoietic Stem Cell Transplantation
Acronym: EVaxAll
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other); University Hospital, Clermont-Ferrand (Other); University Hospital of Saint-Etienne (Other); Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 38RC17.191
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Haemopoietic Stem Cell Transplantation; Allograft
Keywords: haemopoietic stem cell transplantation; vaccine; diphteria; tetanus; haemophilus influenza; poliomyelitis; hepatitis B
MeSH Terms: conditions — Tetanus; Poliomyelitis; Hepatitis B

STUDY DESIGN:
Intervention Model Description: randomized, open-label, prospective, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- good resp. after 3 vacc. inject. (No Intervention): no randomization for a 4th dose.
- bad resp. after 3 vacc. inj., 4th inj (Experimental): After randomization, these patients will receive a 4th dose one month after the 3rd dose.
  Interventions: Drug: 4th dose of hexavalent vaccine 1 month after the 3rd dose
- bad resp. after 3 vacc. inj., no 4th inj (No Intervention): After randomization, these patients will not receive a 4th dose one month after the 3rd dose.

INTERVENTIONS:
Drug: 4th dose of hexavalent vaccine 1 month after the 3rd dose — 4th dose of hexavalent vaccine 1 month after the 3rd dose
  Arms: bad resp. after 3 vacc. inj., 4th inj

SUMMARY:
It is recommended for patients who underwent an hematopoietic stem cell transplantation to receive 6 months after the graft 3 injections of hexavalent vaccine (diphteria-tetanus- poliomyelitis-pertussis-Hib-HBV) within 2 months followed by a booster dose one month after. The patients included in the study will have a measure of their antibody level against 5 pathogens (diphteria toxin, tetanus toxin, Haemophilus influenza b, hepatitis B virus, poliomyelitis virus) one month after the 3rd injection of hexavalent vaccine. If the antibody response is not sufficient, they will be randomized for a 4th dose in the following month. The antibody response will be again measured one month after the 1 year booster dose.

DETAILED DESCRIPTION:
It is recommended for patients who underwent an hematopoietic stem cell transplantation to receive, 6 months after the graft, 3 injections of hexavalent vaccine (diphteria-tetanus- poliomyelitis-pertussis-Hib-HBV) within 2 months, followed by a booster dose one yrar after. However, this strategy do not constantly lead to efficient antibody levels.

the investigators aim to determine whether a 4th dose in the initial vaccine schedule (month 0, 1, 2, and 3) allows to obtain a better response.

After informed consent, the investigators will recruit 6 months after the graft 200 patients who had received an hematopoietic stem cell transplantation . The participants will have a measure of their antibody level against 5 pathogens (diphteria toxin, tetanus toxin, Haemophilus influenza b, hepatitis B virus, poliomyelitis virus) at month 0 (before the 1st hexavalent vaccine injection), and one month after the 3rd injection of this vaccine. If the antibody response is not sufficient, they will be randomized for a 4th dose in the following month.

The one year booster dose will be then injected to all participants, and the antibody response will be again measured one month after this dose. The primary endpoint is to compare the antibody levels at this date in patients who had an unsufficient immune response after the 3rd dose and who received or not a 4rth dose in the initial vaccine schedule.

ELIGIBILITY:
Inclusion Criteria:

* having received an HSTC 6 months before (not more than 2 years)
* not receiving immunosuppressive therapy at inclusion

Exclusion Criteria:

* having received an HSTC 6 months more than 2 years before
* receiving immunosuppressive therapy at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
antibody response 1 month after the one year booster dose | 1 month after the one year booster dose
  antibody level against 5 pathogens (diphteria toxin, tetanus toxin, Haemophilus influenza b, hepatitis B virus, poliomyelitis virus) one month after the 3rd injection of hexavalent vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Olivier EPAULARD, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Epaulard O, Carre M, Hermet E, Corbin V, Tavernier E, Botelho-Nevers E, Daguindau E, Brunel AS, Rohrlich PS, Risso K, Gallet S, Gonnet N, Touati S, Manceau M, Thiebault A. Antibody response to tetanus, diphtheria, poliomyelitis, hepatitis B, and H. influenzae b vaccines in allogeneic hematopoietic stem cell transplant adult recipients: A multicenter trial. PLoS One. 2025 Oct 27;20(10):e0335224. doi: 10.1371/journal.pone.0335224. eCollection 2025. PMID 41144397